CLINICAL TRIAL: NCT01488019
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of Long-Term Use of Perforomist® (Formoterol Fumarate) Inhalation Solution in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study to Evaluate the Safety of Long-Term Use of Perforomist® (Formoterol Fumarate)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201-085
Record Dates: First submitted 2011-11-29; First posted 2011-12-08 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perforomist, nebulization, COPD (Experimental): Active
  Interventions: Drug: Perforomist, nebulization, COPD
- Perforomist-Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Perforomist-Placebo

INTERVENTIONS:
Drug: Perforomist-Placebo — Placebo vehicle, 2mL, twice daily for 52 weeks
  Other Names: Perforomist
  Arms: Perforomist-Placebo
Drug: Perforomist, nebulization, COPD — Perforomist, 20 mcg/2 mL, twice daily for 52 weeks
  Other Names: Formoterol fumarate
  Arms: Perforomist, nebulization, COPD

SUMMARY:
This study is a multi-center, randomized, placebo-controlled study to evaluate the long-term safety of Perforomist® inhalation therapy in subjects with Chronic Obstructive Pulmonary Disease (COPD). Individual participation is approximately 54 weeks, including 52 weeks of double-blind treatment.

DETAILED DESCRIPTION:
None provided.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study requirements, provide written informed consent, and agree to abide by the study protocol and its restrictions
2. Male and female subjects at least 40 years of age with a medical diagnosis of COPD (i.e. persistent presence of dyspnea, cough or sputum production and a history of exposure to risk factors for the disease, such as tobacco smoke)
3. A current or prior history of at least 10 pack-years of cigarette smoking and a baseline breathlessness severity grade of >=2 (Modified Medical Research Council [MMRC] Dyspnea Scale Score) at randomization.
4. Women of child-bearing potential (WOCBP) must have a negative pregnancy test at the screening visit and agree to avoid becoming pregnant for the duration of study by using adequate contraception at study entry and throughout the trial. WOCBP will be advised to notify the Investigator of any change in their pregnancy status. WOCBP include: any female who has experienced menarche and is not post-menopausal (defined as amenorrhea for at least 12 consecutive months), or has not undergone surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation). Women who are using acceptable contraceptive medications or devices to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy) will be considered WOCBP.
5. Able to complete all aspects of the study through the end of the study, including all visits and tests, and self-administration of study medications.

Exclusion Criteria:

1. A medical diagnosis of asthma. Indication of a past history of asthma that is deemed inaccurate to a subject's current condition by the Investigator must be adequately addressed in the medical history.
2. Clinically significant abnormal chest x-ray (CXR) (within the past 12 months) diagnostic of active/significant disease other than COPD.
3. Evidence of any unstable or clinically significant hematopoietic, malignant, cardiovascular, hepatic, renal, neurologic, psychiatric, autoimmune disorder, or condition or disease other than COPD that, in the opinion of the Investigator, could place the subject at increased risk of complications, interfere with study participation, or confound any of the study objectives.
4. Subjects who had radiation or chemotherapy within the previous 12 months.
5. An abnormal laboratory test at screening deemed clinically significant and exclusionary by the Investigator.
6. A history of hypersensitivity to study drugs or their components, including albuterol rescue.

   -

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1071 (Actual)
Dates: Start 2012-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dik Ng, Study Director — Mylan Pharma UK Ltd.
Locations (1):
- Chandar Abboy, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Perforomist Inhalation Solution: Active
  Perforomist Inhalation Solution, 20 mcg/2 mL, twice daily nebulization for 52 weeks
- Matching Placebo: Placebo
  Perforomist Matching Placebo: placebo vehicle, 2mL, twice daily nebulization for 52 weeks
Period: Overall Study
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Started | 541 | 530
Completed | 294 | 226
Not Completed | 247 | 304

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- Perforomist Inhalation Solution: Active
  Perforomist Inhalation Solution, 20mcg/2 mL, twice daily nebulization for 52 weeks
- Total: Total of all reporting groups
Arm/Group | Perforomist Inhalation Solution | Matching Placebo | Total
Number analyzed (Participants) | 541 | 530 | 1071
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.01) | 62.5 (9.17) | 62.6 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 267 | 552
  Male | 256 | 263 | 519
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 26 | 55
  Not Hispanic or Latino | 512 | 504 | 1016
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 483 | 478 | 961
  Black or African American | 51 | 46 | 97
  American Indian or Alaska Native | 0 | 2 | 2
  Asian or Pacific Islander | 4 | 1 | 5
  Other | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 541 | 530 | 1071
Screening COPD Severity (GOLD) n (%) [Count of Participants; unit: Participants]
  Moderate (% Predicted FEV1 50 to <80%) | 274 | 273 | 547
  Severe (% Predicted FEV1 30 to <50%) | 261 | 250 | 511
  Very Severe (% Predicted FEV1 <30%) | 3 | 4 | 7
  Not Reported/Unknown | 3 | 3 | 6
Baseline FEV1 [Mean (Standard Deviation); unit: Litres] — Forced expiratory volume in one second Population: Only subjects with data collected and valid measurements included
  Litres
    number analyzed (Participants) | 539 | 526 | 1065
    (all) | 1.2494 (0.47593) | 1.2926 (0.50496) | 1.2707 (0.49073)
Baseline % Predicted FEV1 [Mean (Standard Deviation); unit: %] — Forced expiratory volume in one second, percent of predicted NHANES III reference values Population: Only subjects with data collected and valid measurements included
  %
    number analyzed (Participants) | 539 | 526 | 1065
    (all) | 43.82 (12.646) | 44.89 (13.787) | 44.35 (13.226)
Baseline FVC [Mean (Standard Deviation); unit: Litres] — Forced vital capacity Population: Only subjects with data collected and valid measurements included
  Litres
    number analyzed (Participants) | 539 | 526 | 1065
    (all) | 2.4276 (0.74347) | 2.4740 (0.78394) | 2.451 (0.76373)
Baseline IC [Mean (Standard Deviation); unit: Litres] — Inspiratory Capacity Population: Only subjects with data collected and valid measurements included
  Litres
    number analyzed (Participants) | 522 | 514 | 1036
    (all) | 1.9458 (0.66598) | 1.9783 (0.66897) | 1.9619 (0.66734)
Number of Pack Years [Mean (Standard Deviation); unit: Pack Years] | 48.37 (26.176) | 50.87 (27.912) | 49.60 (27.066)
Number of Pack Years [Median (Full Range); unit: Pack Years] | 41 [10.0 to 184.0] | 44.00 [10.0 to 232.0] | 43.00 [10.0 to 232.0]
Smoking Status n (%) [Count of Participants; unit: Participants]
  Ex-smoker | 259 | 252 | 511
  Current Smoker | 282 | 278 | 560
Baseline Saint Georges Respiratory Questionnaire Score [Mean (Standard Deviation); unit: units on a scale] — Saint Georges Respiratory Questionnaire comprises 50 items in 3 sections (Symptoms, Activity, Impact) measuring health status in chronic airflow limitation. Symptoms captures level of symptomatology. Activity and Impact responses are either "yes" or "no". Scoring is from 0 to 100; 0 = no life quality impairment. A summary score for all items is calculated and ranges from 0 to 100, where 0 indicates best possible health status, 100 represents worst possible health status. Scores are calculated using weights attached to each item in the questionnaire - 4 unit changes are clinically meaningful. Population: Only subjects with data collected and valid measurements included
  units on a scale
    number analyzed (Participants) | 536 | 529 | 1065
    (all) | 53.429 (16.9607) | 52.550 (16.9953) | 52.992 (16.9756)
Baseline Dyspnea Index [Mean (Standard Deviation); unit: units on a scale] — The Baseline Dyspnea Index (BDI) is an interviewer-administered rating of severity of dyspnea at baseline. It has 3 components: functional impairment, magnitude of task, and magnitude of effort, and each component is rated on a graded scale from 0 (very severe) to 4 (no impairment). The 3 components are summed to provide a total score ranging from 0 to 12. The lower the score, the worse the severity of dyspnea. Population: Only subjects with data collected and valid measurements included
  units on a scale
    number analyzed (Participants) | 539 | 528 | 1067
    (all) | 6.1 (1.99) | 6.2 (1.99) | 6.2 (1.99)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Primary Event of Respiratory Death, First COPD-Related Emergency Room Visit, or First COPD Exacerbation-Related Hospitalisation
Description: The primary endpoint was the combined incidence of respiratory death, first COPD-related ER visit or first COPD exacerbation-related hospitalization (whichever occurred first from the time of randomization to the end of the study). The time-to-first event was measured and analyzed in units of weeks and was summarized by treatment for subjects in the Safety Set. An independent Mortality Adjudication Board was used to evaluate all deaths that occurred in the study and for assigning cause of death and COPD-relatedness.
Time Frame: 0 to 52 weeks
Population: Safety Set - All subjects who were randomized to treatment and took at least one dose of study medication. Subjects were analyzed according to the actual treatment they received for the majority of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Participants | 64 | 57
Statistical Analysis 1: Comparison: Perforomist Inhalation Solution vs Matching Placebo; Test type: Non-Inferiority — The hazard ratio and 90% two-sided confidence interval for the hazard ratio comparing Perforomist to placebo were estimated. Non-inferiority was declared if the upper limit of the two-sided 90% confidence interval was wholly less than 1.5; Regression, Cox — Hazard Ratio was calculated as Perforomist vs Placebo. The non-inferiority margin for the hazard ratio is 1.5. Subjects with no primary event at withdrawal or study completion were treated as censored observations at time of withdrawal; Treatment, site group, and bronchodilator reversibility included as covariates in the model; Hazard Ratio (HR) = 0.965, 90% CI 2-sided [0.711 to 1.308] — Hazard Ratio was calculated as Perforomist Inhalation Solution vs Placebo. The non-inferiority margin for the hazard ratio is 1.5

2. Primary Outcome: Kaplan-Meier Probability of Respiratory Death, First COPD-Related Emergency Room Visit, or First COPD Exacerbation-Related Hospitalisation at 52 Weeks
Description: as for outcome 1
Time Frame: 0 to 52 weeks
Population: as for outcome 1
Measure: Number; unit: percent
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
percent | 15.5 | 14.9

3. Secondary Outcome: Summary of All Cause Mortality, COPD Related Mortality and Respiratory Related Mortality
Description: An independent Mortality Adjudication Board was used to evaluate all deaths that occurred in the study and for assigning cause of death and COPD-relatedness.
Time Frame: 0 to 52 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Participants
  Incidence of All Cause Mortalities | 3 | 10
  Incidence of Respiratory Related Mortalities | 0 | 1
  Incidence of COPD Related Mortalities | 0 | 1

4. Secondary Outcome: Individual Components of the Primary Composite Endpoint - First COPD-related ER Visit and First COPD Exacerbation-Related Hospitalization
Time Frame: 0 to 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Participants
  Subjects with a COPD- related ER Visit | 46 | 47
  Subjects with a COPD-Related Hospitalization | 39 | 43

5. Secondary Outcome: Number of Subjects With Protocol-Defined COPD Exacerbation
Description: COPD exacerbations were defined as events in the natural course of disease characterized by an increase from baseline in two of the following symptoms: dyspnea, cough, and sputum production that was beyond normal day-to-day variations, was acute in onset, that persisted for at least two consecutive days, and that warranted a change in their regular medication. The change could be either the initiation of additional treatment(s) or the intensification of a treatment the subject was already receiving, and the change must have been specifically to address the exacerbation event. COPD exacerbations occurring after the time of withdrawal or completion of the study were not included.
Time Frame: 0 to 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Participants | 142 | 135

6. Secondary Outcome: Kaplan-Meier Probability of Protocol Defined COPD Exacerbation at 52 Weeks
Description: COPD exacerbations were defined as events in the natural course of disease characterized by an increase from baseline in two of the following symptoms: dyspnea, cough, and sputum production that was beyond normal day-to-day variations, was acute in onset, that persisted for at least two consecutive days, and that warranted a change in their regular medication.The change could be either the initiation of additional treatment(s) or the intensification of a treatment the subject was already receiving, and the change must have been specifically to address the exacerbation event. COPD exacerbations occurring after the time of withdrawal or completion of the study were not included.
Time Frame: 0 to 52 weeks
Population: as for outcome 1
Measure: Number; unit: percent
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
percent | 34.7 | 34.0

7. Secondary Outcome: FEV1 Changes From Baseline at Months 3, 6, 9 and 12
Time Frame: On treatment at months 3, 6, 9 and 12
Population: Full Analysis Set: all subjects randomized who took at least one dose of study medication. Subjects were analyzed according to their assigned treatment at randomization. Only subjects with data collected and valid measurements included
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Litres
  Change from Baseline FEV1: Month 3: number analyzed (Participants) | 486 | 435
  Change from Baseline FEV1: Month 3 | 0.058 (0.0116) | 0.016 (0.0123)
  Change from Baseline FEV1: Month 6: number analyzed (Participants) | 366 | 293
  Change from Baseline FEV1: Month 6 | 0.057 (0.0130) | 0.017 (0.0143)
  Change from Baseline FEV1: Month 9: number analyzed (Participants) | 314 | 250
  Change from Baseline FEV1: Month 9 | 0.050 (0.0136) | 0.029 (0.0151)
  Change from Baseline FEV1: Month 12: number analyzed (Participants) | 294 | 227
  Change from Baseline FEV1: Month 12 | 0.030 (0.0144) | 0.000 (0.0160)

8. Secondary Outcome: FVC Changes From Baseline at Months 3, 6, 9 and 12
Time Frame: On treatment at months 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Litres
  Change from Baseline FVC: Month 3: number analyzed (Participants) | 486 | 435
  Change from Baseline FVC: Month 3 | 0.1051 (0.40479) | 0.0062 (0.38724)
  Change from Baseline FVC: Month 6: number analyzed (Participants) | 366 | 293
  Change from Baseline FVC: Month 6 | 0.1006 (0.38875) | -0.0241 (0.37124)
  Change from Baseline FVC: Month 9: number analyzed (Participants) | 314 | 250
  Change from Baseline FVC: Month 9 | 0.1009 (0.39533) | -0.0254 (0.40947)
  Change from Baseline FVC: Month 12: number analyzed (Participants) | 294 | 227
  Change from Baseline FVC: Month 12 | 0.0645 (0.43490) | -0.0581 (0.38069)

9. Secondary Outcome: IC Changes From Baseline at Months 3, 6, 9 and 12
Time Frame: On treatment at months 3, 6, 9 and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Litres
  Change from Baseline IC: Month 3: number analyzed (Participants) | 467 | 420
  Change from Baseline IC: Month 3 | 0.0287 (0.42478) | -0.0119 (0.39505)
  Change from Baseline IC: Month 6: number analyzed (Participants) | 354 | 287
  Change from Baseline IC: Month 6 | 0.0440 (0.44862) | -0.0106 (0.43483)
  Change from Baseline IC: Month 9: number analyzed (Participants) | 306 | 247
  Change from Baseline IC: Month 9 | 0.1584 (1.84290) | -0.0118 (0.43513)
  Change from Baseline IC: Month 12: number analyzed (Participants) | 284 | 221
  Change from Baseline IC: Month 12 | 0.0477 (0.48057) | -0.0105 (0.44289)

10. Secondary Outcome: Saint Georges Respiratory Questionnaire Scores: Changes From Baseline at Months 3, 6, 9, 12
Description: Saint Georges Respiratory Questionnaire comprises 50 items in 3 sections, Symptoms, Activity, Impact, measuring health status in chronic airflow limitation. Symptoms captures level of symptomatology. Activity and Impact responses are either "yes" or "no". Scoring is from 0 to 100; 0 = no life quality impairment. A summary score for all items is calculated and ranges from 0 to 100, where 0 indicates best possible health status, 100 represents worst possible health status. Scores are calculated using weights attached to each item in the questionnaire - 4 unit changes are clinically meaningful.
Time Frame: On treatment at months 3, 6, 9 and 12
Population: Full Analysis Set: all subjects randomized who took at least one dose of study medication. Subjects were analyzed according to their assigned treatment at randomization. Only subjects with data collected were included
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
units on a scale
  Change from Baseline SGRQ Total Score: Month 3: number analyzed (Participants) | 502 | 465
  Change from Baseline SGRQ Total Score: Month 3 | -3.252 (0.5472) | -2.027 (0.5727)
  Change from Baseline SGRQ Total Score: Month 6: number analyzed (Participants) | 377 | 299
  Change from Baseline SGRQ Total Score: Month 6 | -2.329 (0.6541) | -2.511 (0.7156)
  Change from Baseline SGRQ Total Score: Month 9: number analyzed (Participants) | 315 | 255
  Change from Baseline SGRQ Total Score: Month 9 | -2.021 (0.7022) | -2.115 (0.7681)
  Change from Baseline SGRQ Total Score: Month 12: number analyzed (Participants) | 294 | 231
  Change from Baseline SGRQ Total Score: Month 12 | -1.453 (0.7559) | -1.475 (0.8345)

11. Secondary Outcome: Transition Dyspnea Index
Description: The Transition Dyspnea Index (TDI) measures changes in dyspnea severity from the baseline as established by the BDI. It has 3 components: change in functional impairment, change in magnitude of task, and change in magnitude of effort, and each component is rated on a scale ranging from -3 (major deterioration) to +3 (major improvement). The 3 components are summed to provide a total score ranging from -9 to +9. The lower the score, the more deterioration in severity of dyspnea.
Time Frame: On treatment at months 3, 6, 9 and 12
Population: Full Analysis Set: all subjects randomized who took at least one dose of study medication. Subjects were analyzed according to their assigned treatment at randomization.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Perforomist Inhalation Solution: Active
  Perforomist, nebulization, COPD: Perforomist, 20 mcg/2 mL, twice daily for 52 weeks
- Matching Placebo: Placebo
  Perforomist-Placebo: Placebo vehicle, 2mL, twice daily for 52 weeks
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
units on a scale
  Month 3: number analyzed (Participants) | 508 | 464
  Month 3 | 0.7 (0.11) | 0.0 (0.12)
  Month 6: number analyzed (Participants) | 380 | 298
  Month 6 | 0.5 (0.13) | 0.4 (0.14)
  Month 9: number analyzed (Participants) | 320 | 255
  Month 9 | 0.7 (0.14) | 0.4 (0.15)
  Month 12: number analyzed (Participants) | 297 | 231
  Month 12 | 0.5 (0.14) | 0.6 (0.16)

12. Secondary Outcome: Health Care Utilization and Economic Impact - Number of Emergency Department Visits
Time Frame: 0 to 52 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Participants
  0 | 447 | 437
  1 | 78 | 75
  2 | 15 | 16
  >=3 | 1 | 2

13. Secondary Outcome: Summary of Subjects Requiring Intubation or Non-Invasive Ventilation
Time Frame: 0 to 52 weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Participants | 3 | 10

14. Secondary Outcome: Rescue Medication Usage
Description: Number of puffs of rescue medication (albuterol pMDI) used per day
Time Frame: 0 to 52 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Mean Puffs per Day
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
Number analyzed (Participants) | 541 | 530
Mean Puffs per Day
  Baseline: number analyzed (Participants) | 530 | 515
  Baseline | 2.55 (2.496) | 2.52 (2.484)
  Treatment Phase: number analyzed (Participants) | 478 | 455
  Treatment Phase | 1.92 (2.063) | 2.35 (2.521)

ADVERSE EVENTS:
Time Frame: Approximately 14 months (date of signature of the Informed Consent Form to 30 days after last dose of study drug)
Description: Subject Deaths during the Study:
  Perforomist x3 (Neoplasms x2, Cardiac Disorders x1) Placebo x10 (Respiratory, Thoracic and Mediastinal Disorders x1, Neoplasms x2, Cardiac Disorders x5, Infections and Infestations x1, Injury x1)
Arm/Group | Perforomist Inhalation Solution | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 3/541 | 10/530
Serious Adverse Events (participants affected / at risk) | 86/541 | 85/530
Other Adverse Events (participants affected / at risk) | 374/541 | 369/530
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perforomist Inhalation Solution (N=541) | Matching Placebo (N=530)
COPD (Respiratory, thoracic and mediastinal disorders) | 39 | 40
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Acute Myocardial Infarction (Cardiac disorders) | 2 | 6
Pneumonia (Infections and infestations) | 10 | 10
Lobar Pneumonia (Infections and infestations) | 2 | 6
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 3
Atrial fibrillation (Cardiac disorders) | 2 | 2
Cardiac arrest (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Papilloedema (Eye disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 3
Non-cardiac chest pain (General disorders) | 2 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Sepsis (Infections and infestations) | 2 | 4
Influenza (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 0 | 3
Bronchitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchitis pneumococcal (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gallbladder abscess (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 1 | 3
Thalamic infarction (Nervous system disorders) | 0 | 2
Basal ganglia infarction (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Alcohol abuse (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 4
Renal failure (Renal and urinary disorders) | 2 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Penile necrosis (Reproductive system and breast disorders) | 0 | 1
Priapism (Reproductive system and breast disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perforomist Inhalation Solution (N=541) | Matching Placebo (N=530)
Upper Respiratory Tract Infection (Infections and infestations) | 36 | 32
Bronchitis (Infections and infestations) | 34 | 26
COPD (Respiratory, thoracic and mediastinal disorders) | 164 | 145
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 35 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 24
Nausea (Gastrointestinal disorders) | 18 | 7
Diarrhea (Gastrointestinal disorders) | 13 | 11
Constipation (Gastrointestinal disorders) | 11 | 6
Nasopharyngitis (Infections and infestations) | 24 | 18
Sinusitis (Infections and infestations) | 25 | 12
Pneumonia (Infections and infestations) | 18 | 18
Urinary Tract Infection (Infections and infestations) | 14 | 13
Influenza (Infections and infestations) | 11 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 12 | 9
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 12 | 8
Headache (Nervous system disorders) | 21 | 22
Anxiety (Psychiatric disorders) | 12 | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Hypertension (Vascular disorders) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes